CLINICAL TRIAL: NCT00783653
Title: Phase I/II Clinical Study of SU11248 (Sutent) Combined With Standard Chemotherapy With Cytosine Arabinoside and Daunorubicin in Patients With FLT3 Mutated AML Over 60 Years of Age
Brief Title: Clinical Study of SU 11248 (Sutent) Combined With Standard Chemotherapy in Patients With FLT3 Mutated AML Over 60 Years
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG 10/07; AMLSG-SU11248
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; FLT3; acute myeloid leukemia; FLT 3 inhibitor; FLT3 mutated AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sunitinib — 25 mg or 37,5 mg daily dose until DLT
  Other Names: SU11248, Sutent

SUMMARY:
In this study safety and tolerability of two dose levels of SU 11248 (sutent) with standard chemotherapy in patients with FLT3 mutated AML over 60 years will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary or secondary acute myeloid leukemia (any FAB type, except M3).
* No prior systemic chemotherapy for AML except hydroxyurea. Cytoreductive therapy with hydroxyurea is recommended if WBC is > 50.000/µl, but should cease at least one day prior to starting study medication
* Patient age equal or of greater than 60 years
* Patients must have FLT3 mutated AML, either ITD or kinase domain mutations
* ECOG Performance score 3 or less (Karnofsky Performance Score >40%).
* Life expectancy more than four weeks.
* Adequate hepatic and renal function, as defined by serum transaminases <2.5x ULN, bilirubin <1.5x ULN. Creatinine <1.5x ULN.
* Patients must provide written informed consent to participate in the trial.
* Normal heart function on cardiac ultrasound
* Prothrombin time (PT) and partial thromboplastin time (PTT) <=1.5 x ULN
* Serum albumin >=3.0 g/dl
* Serum amylase and lipase <=1.0 x ULN
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment:

* Treatment with any investigational agent within four weeks.
* Known HIV infection
* Presence of any medical or psychiatric condition which may limit full compliance with the study, including but not limited to:
* Presence of CNS leukaemia
* Unresolved toxicity from previous anti-cancer therapy or incomplete recovery from surgery.
* Any of the following within the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or other thromboembolic event.
* Current treatment with therapeutic doses of anticoagulant (low dose Coumadin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
* Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy).
* Pre existing thyroid abnormality of thyroid function that cannot be maintained in the normal range with medication.
* Ongoing cardiac dysrhythmias of NCI CTCAE Grade >=2, atrial fibrillation of any Grade, or prolongation of the QTc interval to >450 msec for males or >470 msec for females.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Definition of a recommended Phase III dose and determination CTC version 3.0 grade 3-5 non-hematological toxicities of SU11248 in combination with standard induction and consolidation chemotherapy | April 2011

SECONDARY OUTCOMES:
Overall safety profile of SU11248 characterized by type, frequency, severity (graded using NCI CTCAE Version 3.0), timing and relatedness of adverse events (AEs) and laboratory | April 2011
Objective tumor response, as defined using the revised recommendations of the International Working Group for diagnosis, standardization of response criteria in Acute Myeloid Leukemia for AML | April 2011

CONTACTS AND LOCATIONS:
Overall Officials: Walter Fiedler, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (5):
- Germany (5):
  - Prof. Dr. med. Walter Fiedler, Hamburg
  - PD Dr. med. Jürgen Krauter, Hanover
  - Dr. Katharina Götze, München
  - Prof. Dr. Helmut R. Salih, Tübingen
  - Dr. Richard Schlenk, Ulm

REFERENCES:
- [Result] Fiedler W, Kayser S, Kebenko M, Janning M, Krauter J, Schittenhelm M, Gotze K, Weber D, Gohring G, Teleanu V, Thol F, Heuser M, Dohner K, Ganser A, Dohner H, Schlenk RF. A phase I/II study of sunitinib and intensive chemotherapy in patients over 60 years of age with acute myeloid leukaemia and activating FLT3 mutations. Br J Haematol. 2015 Jun;169(5):694-700. doi: 10.1111/bjh.13353. Epub 2015 Mar 29. PMID 25818407